CLINICAL TRIAL: NCT06699095
Title: "Tele-riabilitazione in Sclerosi Multipla: Continuità Terapeutica Domiciliare Dopo Trattamento Di Neuro-riabilitazione Intensiva, Studio Randomizzato Controllato Con Piattaforma Integrata Per La Riabilitazione Del Disequilibrio"
Brief Title: Home Rehabilitation As Continuity of Care in MS
Acronym: HoReConCareMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Istituto Auxologico Italiano (Other); Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HoReConCareMS
Record Dates: First submitted 2024-11-12; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
Keywords: Balance rehabilitation; Telemedicine; Home rehabilitation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional, telemedicine group (Experimental): Patients will perform a 12 weeks rehabilitation program through telemedicine at home after intensive rehabilitation in hospital
  Interventions: Device: Telerehabilitation
- Control group (No Intervention): Patients will perform a 12 weeks maintenance rehabilitation program as usual care (TAU treatment as usual) at home after intensive rehabilitation in hospital

INTERVENTIONS:
Device: Telerehabilitation — Patients will perform a 12 weeks rehabilitation program through telemedicine at home after intensive rehabilitation in hospital. Balance rehabilitation program will be scheduled on the patients' need and ability to be performed three times a week with high levels of satisfaction and safety at home under remote control of the physical therapist.
  Other Names: Telemedicine
  Arms: Interventional, telemedicine group

SUMMARY:
RCT pilot study to evaluate adherence, satisfaction and feasibility in the use of a telemedicine station for balance rehabilitation in patients with multiple sclerosis.

The platform is designed as a tool for maintenance rehabilitation in a home setting and not as an alternative to intensive treatment in hospital, and is therefore compared to maintenance treatment as usual (TAU) after intensive treatment.

DETAILED DESCRIPTION:
Balance deficit represents one of the most frequent symptoms in patients with Multiple Sclerosis (PwMS) and one of the most disabling. Neuromotor rehabilitation is a fundamental tool for managing these symptoms: therapeutic exercise is currently the best choice for treating balance deficit. Once improvements has been achieved, this generally does not persist for a long time due to the underlying chronic-degenerative pathology: this reduction in clinical benefit, which can be graphically defined as a 'loss curve', is difficult to define due to individual differences, but it affects all MS patients. In recent years, new technologies are emerging, such as virtual reality and serious gaming, which are not presented as an alternative to intensive treatment but could find their ideal dimension in extensive treatment, allowing the patient to maintain the results achieved once the period of intensive treatment in a specialised rehabilitation facility is over. The specific objectives of this feasibility study are: to refine technical aspects of the Neuro Rehability system, to evaluate acceptability and satisfaction with its use by PwMS, to evaluate the recruitment process, adherence to the intervention, the number of drop-outs and identify potential problems, to evaluate the human resource requirements for the subsequent RCT study, to estimate the intervention effect and its variance necessary to calculate the appropriate sample size for the RCT.. Assessments will be carried out before the start (T0) and at the end (T1) of the treatment. The control group is asked to continue performing at home the normal physical activities that they may already be performing for the duration of the 12 weeks (TAU = treatment as usual). The experimental group is asked to perform the exercises of the Rehability platform, previously set up by the rehabilitation team on the basis of the training performed during the intensive rehabilitation period in the facility, at least 3 times a week and for at least 40 minutes per session. For both groups, no rehabilitation treatment will be possible except sphincter and phoniatric rehabilitation and psychological support. A descriptive statistical analysis will be used to describe the demographic and clinical characteristics of the sample. Standard data analysis techniques will be used to analyse the variables collected in both the feasibility study and the RCT. An electronic CRF will be set up to collect: clinical and demographic data on the recruited subjects; results of the tests/questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale score between 3 and 6
* Sensory Organisation Test Equitest values indicating balance impairment

Exclusion Criteria:

* visual impairments
* orthopedic impairments
* inability to perform balance rehabilitation in stand up position

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-11-06 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Home rehabilitation, from the end of the intensive treatment to the follow up evaluation (12 weeks)
  Safety in the use of the telemedicine system - number of sessions played and number of adverse events/number of dropouts

SECONDARY OUTCOMES:
Telehealthcare Satisfaction Questionnaire (TSQ) | From the end of the intensive treatment to the follow up evaluation (12 weeks)
  Satisfaction levels perceived by patients in the use of the telemedicine system evaluating benefit, usability, self-concept, privacy, quality of life, comfort. Scores go from zero to 4 (zero is equivalent to minimum benefit in using the telemedicine system, 4 is equivalent to maximum benefit).
Telehealthcare Usability Questionnaire (TUQ) | From the end of the intensive treatment to the follow up evaluation (12 weeks)
  Satisfaction levels perceived by operators in the use of the telemedicine system evaluating twenty-one items about the usability of the system. Scores evaluate the level of agreement with statements about the system and go from zero (totally disagree) to 7 (totally agree).
Timed Up and Go test (TUG) | From the end of the intensive treatment to the follow up evaluation (12 weeks)
  Pre and post intervention assessment of mobility, balance, walking ability, and fall risk. Patients have to complete a sit to stand from a set chair and walk for 7 meters, turn around and sit down again, the score is the time needed to complete the test (seconds).
Timed 10-Meter Walk Test | From the end of the intensive treatment to the follow up evaluation (12 weeks)
  Pre and post intervention assessment of walking ability in terms of time (seconds) and steps necessary to complete a 10 meters path.
Equiscale test | From the end of the intensive treatment to the follow up evaluation (12 weeks)
  Pre and post intervention assessment of balance. Patients have to complete eight items evaluation static and dynamic balance (i.e. sit to stand, stand still with open and closed eyes) with a score from zero to 2 (zero is considered as not able to complete, 1 is partially able, 2 is totally able), total score is 16 points.
12-Item Multiple Sclerosis Walking Scale | From the end of the intensive treatment to the follow up evaluation (12 weeks)
  The 12-item Multiple Sclerosis Walking Scale (MSWS-12) is a self-report measure of the impact of MS on the individual's walking ability. The scoring provides options 1-5 for each item, with 1 meaning no limitation and 5 meaning extreme limitation on the gait-related item. Total score is 60. Final score is calculated as a percentage of walking impairment (score x 100/60).
Multiple Sclerosis Quality of Life Questionnaire-54 (MSQoL-54) | From the end of the intensive treatment to the follow up evaluation (12 weeks)
  The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The summary scores are the physical health composite summary and the mental health composite summary.
  Multiple Sclerosis Quality of Life-54 (MSQOL-54) There is no single overall score for the MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores.
Modified Fatigue Impact Scale (M-FIS) | From the end of the intensive treatment to the follow up evaluation (12 weeks)
  The MFIS is a modified form of the Fatigue Impact Scale based on items derived from interviews with MS patients concerning how fatigue impacts their lives.
  Scoring the MFIS Items on the MFIS can be aggregated into three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities.
  Physical Subscale can range from 0 to 36. It is computed by adding raw scores on the following items: 4+6+7+10+13+14+17+20+21.
  Cognitive Subscale can range from 0 to 40. It is computed by adding raw scores on the following items: 1+2+3+5+11+12+15+16+18+19.
  Psychosocial Subscale can range from 0 to 8. It is computed by adding raw scores on the following items: 8+9.
  Total MFIS Score The total MFIS score can range from 0 to 84. It is computed by adding scores on the physical, cognitive, and psychosocial subscales.
Patient Health Engagement scale (PHE scale) | From the end of the intensive treatment to the follow up evaluation (12 weeks)
  The Patient Health Engagement Model (PHE Model) is a psychological engagement model that allows to diagnose and study the experience of active engagement of patients in its prevention and treatment pathway.
  Scoring is referred to five statements about the engagement level of the patient. Scores go from zero (less level of engagment) to 7 (higher level of engagement) and the total score is 35.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Istituto Auxologico Italiano, Milan, MI
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, MI
  - IRCCS Santa Maria nascente - Fondazione Don Gnocchi, Milan, MI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benzel E. Empowerment. World Neurosurg. 2022 Jan;157:xv. doi: 10.1016/j.wneu.2021.10.132. No abstract available. PMID 34929787
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Truijen S, Abdullahi A, Bijsterbosch D, van Zoest E, Conijn M, Wang Y, Struyf N, Saeys W. Effect of home-based virtual reality training and telerehabilitation on balance in individuals with Parkinson disease, multiple sclerosis, and stroke: a systematic review and meta-analysis. Neurol Sci. 2022 May;43(5):2995-3006. doi: 10.1007/s10072-021-05855-2. Epub 2022 Feb 17. PMID 35175439
- [Background] Yazgan YZ, Tarakci E, Tarakci D, Ozdincler AR, Kurtuncu M. Comparison of the effects of two different exergaming systems on balance, functionality, fatigue, and quality of life in people with multiple sclerosis: A randomized controlled trial. Mult Scler Relat Disord. 2020 Apr;39:101902. doi: 10.1016/j.msard.2019.101902. Epub 2019 Dec 21. PMID 31924591
- [Background] Cimino V, Chisari CG, Raciti G, Russo A, Veca D, Zagari F, Calabro RS, Patti F. Objective evaluation of Nintendo Wii Fit Plus balance program training on postural stability in Multiple Sclerosis patients: a pilot study. Int J Rehabil Res. 2020 Sep;43(3):199-205. doi: 10.1097/MRR.0000000000000408. PMID 32371848
- [Background] Celesti A, Cimino V, Naro A, Portaro S, Fazio M, Villari M, Calabro RS. Recent Considerations on Gaming Console Based Training for Multiple Sclerosis Rehabilitation. Med Sci (Basel). 2022 Feb 11;10(1):13. doi: 10.3390/medsci10010013. PMID 35225946
- [Background] Kim Y, Lai B, Mehta T, Thirumalai M, Padalabalanarayanan S, Rimmer JH, Motl RW. Exercise Training Guidelines for Multiple Sclerosis, Stroke, and Parkinson Disease: Rapid Review and Synthesis. Am J Phys Med Rehabil. 2019 Jul;98(7):613-621. doi: 10.1097/PHM.0000000000001174. PMID 30844920
- [Background] Garcia-Munoz C, Cortes-Vega MD, Heredia-Rizo AM, Martin-Valero R, Garcia-Bernal MI, Casuso-Holgado MJ. Effectiveness of Vestibular Training for Balance and Dizziness Rehabilitation in People with Multiple Sclerosis: A Systematic Review and Meta-Analysis. J Clin Med. 2020 Feb 21;9(2):590. doi: 10.3390/jcm9020590. PMID 32098162
- [Background] Donze C, Massot C. Rehabilitation in multiple sclerosis in 2021. Presse Med. 2021 Jun;50(2):104066. doi: 10.1016/j.lpm.2021.104066. Epub 2021 May 11. PMID 33989721
- [Background] Manjaly ZM, Harrison NA, Critchley HD, Do CT, Stefanics G, Wenderoth N, Lutterotti A, Muller A, Stephan KE. Pathophysiological and cognitive mechanisms of fatigue in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2019 Jun;90(6):642-651. doi: 10.1136/jnnp-2018-320050. Epub 2019 Jan 25. PMID 30683707
- [Background] Cameron MH, Nilsagard Y. Balance, gait, and falls in multiple sclerosis. Handb Clin Neurol. 2018;159:237-250. doi: 10.1016/B978-0-444-63916-5.00015-X. PMID 30482317
- [Background] Berrigan LI, Fisk JD, Patten SB, Tremlett H, Wolfson C, Warren S, Fiest KM, McKay KA, Marrie RA; CIHR Team in the Epidemiology and Impact of Comorbidity on Multiple Sclerosis (ECoMS). Health-related quality of life in multiple sclerosis: Direct and indirect effects of comorbidity. Neurology. 2016 Apr 12;86(15):1417-1424. doi: 10.1212/WNL.0000000000002564. Epub 2016 Mar 9. PMID 26962068
- [Background] Herrera WG. Vestibular and other balance disorders in multiple sclerosis. Differential diagnosis of disequilibrium and topognostic localization. Neurol Clin. 1990 May;8(2):407-20. PMID 2193219